CLINICAL TRIAL: NCT06192862
Title: Effectiveness of Theory-based Outreach Using Mobile Health Technology in Colorectal Cancer Screening Uptake: a Randomized Controlled Trial
Brief Title: Effectiveness of Using Mobile Health Technology in Colorectal Cancer Screening Uptake
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022.614
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: CRC, Colorectal Cancer
Keywords: colorectal cancer, screening, fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient will be randomized into either Text reminder (control) group or Chatbot outreach group
Masking Description: There will no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text reminder group (control) (No Intervention): Randomized subjects to the text reminder group will be asked about their intention to undergo CRC screening in the next 6 months. For those who are at pre-contemplation and contemplation stage, a standard text message will be delivered to invite them to undergo CRC screening by informing them that they are due to CRC screening because they are aged >50 years and are yet to receive CRC screening. No HBM-based health education video or personalized risk assessment will be provided. The chatbot then asks the subject's intention to undergo CRC screening again. For those who propelled to preparation stage or those who are at preparation stage at the beginning, the website link of the government-subsidized CRC screening program which lists the names of all primary care physicians and their contact and co-payment information will be provided.
- Chatbot outreach group (Experimental): Subjects in chatbot outreach group will be asked about their intention to undergo CRC screening in the next 6 months and their TTM stage will be determined according to their answers. For subjects who are at preparation stage, the chatbot will further request for the preferred district to have a consultation under the government-subsidized CRC screening.
  For subjects who are at pre-contemplation stage, the chatbot will deliver an HBM-based health education video filmed by gastroenterologists and colorectal cancer survivor who has been diagnosed by screening. The subject's intention will be asked again after the video.
  For those who upgrade to contemplation stage or remain at pre-contemplation stage and those who are at contemplation stage at the beginning, the chatbot will assess the personalized risk of CRC using the Asia-Pacific Colorectal Screening Score (APCS). Finally, the subject's intention to undergo screening will be asked for the last time.
  Interventions: Behavioral: Assessment of screening intention and Transtheoretical Model stages for CRC screening

INTERVENTIONS:
Behavioral: Assessment of screening intention and Transtheoretical Model stages for CRC screening — Screening Intentions will be measured by asking the subject, ""How much do you agree or disagree: I am intending to have colon cancer screening within the next 6 months". Subjects who "strongly disagrees" or "somewhat disagrees" are considered not having screening intention. Subjects who "somewhat agrees" or "strongly agrees" are considered having screening intention. For subjects who has screening intention, they will be asked if they have plan to arrange a consultation with primary care physician to collect FIT kits in next 3 months.
  Arms: Chatbot outreach group

SUMMARY:
In Hong Kong, Colorectal cancer (CRC) ranked second in both cancer incidence and mortality, accounting for 16.7% of all new cancer cases and 14.6% of all cancer-related deaths in 2019. There was a staggering 2.5-fold increase in the number of newly diagnosed CRC cases from 1584 to 2019.

The fecal immunochemical test (FIT) helps reduce the incidence and mortality of CRC and is widely used for population-based CRC screening. The government-subsidized CRC screening program was launched in Hong Kong as a pilot in 2015 and fully implemented in 2020. The program was subsidized for asymptomatic Hong Kong residents, aged 50-75 years, to receive FIT screening every two years. A subsidized follow-up colonoscopy was offered for a positive FIT result. For a negative FIT result, the participant was advised to repeat the screening two years later.

Despite the subsidy and promotion, the uptake rate of the population-based colorectal cancer screening was low. Only 275,000 (~10%) underwent FIT screening under this program as of 31st December 2021. Efforts have been made to increase the rate. Outreach is the active dissemination of screening outside of the primary care setting, and it also includes mailing, texting, and calling to encourage scheduling of screening procedures.

All eligible subjects will be randomized and allocated to receive either intervention (chatbot) or standard of care (text reminder) in a 1:1 allocation ratio. A fully automated chatbot will be developed and maintained in collaboration with IT experts on the WhatsApp Messenger platform for its wide popularity in local older adults and user-friendly interfaces for extensions. Depending on the randomization group, it delivers either a standard text reminder of CRC screening or health education in text and video formats with a series of questions on personalized risk assessment of CRC and information of primary care physicians under a government-subsidized CRC screening program according to the subject's preferred district. The same professional team will maintain the health status of the chatbot during the intervention period. A monthly review of chatbot performance will be conducted. A feedback loop is also incorporated into the chatbot, and users are invited to leave comments. Accordingly, improvements will be made, and the questions raised by the subjects will be collected and used to construct a data bank for the future development of Artificial intelligence (AI)-enabled chatbots.

DETAILED DESCRIPTION:
It was technically infeasible to conduct fecal test outreach by mailing the test kits in Hong Kong because the government-subsidized colorectal cancer screening program required consultation with a primary care physician to assess the subjects' health condition, and their eligibility before distributing the fecal test kits. Similar to colonoscopy screening outreach, an alternative method is to provide contact information with primary care physicians located in the subject's preferred district via mobile messenger-based chatbots to arrange a consultation for FIT screening. Chatbots have already proven to be useful in increasing the intention to vaccinate against COVID-19.

Moreover, CRC screening uptake is highly associated with Health Belife Model (HBM) constructs and high risk perception of developing CRC is associated with higher screening uptake rate. HBM-based education and Trans-Theoretical Model (TTM)-based personalized risk assessment of CRC may increase the screening uptake rate by improving their knowledge of CRC screening (in terms of susceptivity, perceived benefits, and cues to actions) and informing subjects that they are at a relatively higher risk of developing CRC.

The CRC screening uptake rate in Hong Kong was 10%, and there is no established evidence to increase the uptake rate of FIT screening for CRC by outreach using mobile health technology or psychological theory-based interventions. A theory-based mobile messenger-initiated chatbot is a potential solution to this problem.

---------------

Telephone follow-up

All subjects will be interviewed by phone three and six months after recruitment and asked if they have participated in the government-subsidized CRC screening program and CRC screening completion rate. The date of participation, completion of CRC screening, and FIT results will also be assessed. The reasons for not participating in the CRC screening program will be documented. We will also ask the subjects who have completed CRC screening if our chatbot or text reminder motivated them to uptake or there is exposure to any possible confounders, e.g., community initiative, related symptom onset, healthcare worker advice and family member or friend initiative, etc. A cash coupon of $50 Hong Kong Dollar will be mailed to the subject upon completion of telephone follow-up.

Focus group discussions

12 focus group discussions (6-8 participants per group) will be conducted after the telephone follow-up. The purpose of the focus group discussions is to identify the process factors to understand how the study intervention influence screening uptake behaviors and explore the complexity of FIT screening and reveal, based on the participants' accounts, the barriers, and facilitators for them to uptake FIT screening. Six groups from each RCT arm will be convened. For each discussion session, an experienced moderator from our research team will introduce our study aims, lead the discussion in a semi-structured format based on the discussion protocol, and ask clarifications when necessary. Another assistant will take notes and address contingent issues. Each focus group will be audiotaped and last for 1.5-2.5 hours. All participants will sign a written consent form before the focus group session and will be given some incentives at the end of the session to compensate for their time.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years old
* asymptomatic and eligible to enroll in a government-subsidized colorectal cancer screening program
* subjects themselves or their family members living in the same household with access to WhatsApp Messenger
* able to read Chinese
* willingness to be followed up by telephone

Exclusion Criteria:

* subject without access to WhatsApp Messenger
* unable to provide informed consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
CRC screening uptake rate | during the study period up to six months
  The primary outcome is the CRC screening uptake rate, defined as participation in and completion of the government-subsidized CRC screening program by returning valid FIT kits at three months after intervention and at six months after recruitment

SECONDARY OUTCOMES:
Likert scale | during the study period up to six months
  baseline intention of CRC screening before intervention, measured by 4 point Likert scale (1 = strongly disagree; 2 = somewhat disagree; 3 = somewhat agree and 4 = strongly agree) and the change in screening intent immediately after each intervention, evaluated by calculating point difference between pre- and post-intervention
time interval | during the study period up to six months
  time interval to participate (Date of FIT kits collection minus date of study intervention) and complete screening after recruitment (Date of return of valid FIT kit minus date of study intervention)
qualitative factors checklist associated with CRC screening | during the study period up to six months
  reason for not participating in screening (common local barriers to CRC screening, including, financial difficulty, limited services accessibility, screening-induced bodily discomfort, physical harm, embarrassment, apprehension, time constraints and others) checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Digestive Health, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There will be no plan to share Individual participant data

REFERENCES:
- [Derived] Hu Y, Lau WM, Wang ZJ, Tang RSY, Wu X, Mo PKH, Wong SYS, Meng MLH, Dong D, Sung JJY, Lam TYT. Theory-based chatbot for promoting colorectal cancer screening in a community setting in Hong Kong: study protocol of a randomised controlled trial. BMJ Open. 2025 Jul 10;15(7):e103857. doi: 10.1136/bmjopen-2025-103857. PMID 40639841